CLINICAL TRIAL: NCT05645757
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous Ertapenem in Combination With Zidebactam (WCK 6777) In Healthy Adult Subjects
Brief Title: Safety Study of Intravenous Ertapenem in Combination With Zidebactam (WCK 6777)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-0013
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2022-09-22

CONDITIONS: Bacterial Infection
Keywords: Double-blind; Intravenous Ertapenem; Phase 1; Safety; Zidebactam (WCK 6777)
MeSH Terms: conditions — Bacterial Infections | interventions — Ertapenem; zidebactam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All investigative site personnel, study volunteers, DMID, Wockhardt and DVC personnel will remain blinded through database lock, with the exception of an unblinded pharmacist/verifier at the research site, an unblinded SDCC biostatistician, and a DMID/CMS manager responsible for PK sample storage.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): WCK 6777 (Ertapenem 1 g combined with Zidebactam 1 g) or placebo administered by 100 ml of intravenous infusion (IV) for 30 (±5) minutes once daily for 7 days. N= 8
  Interventions: Drug: Ertapenem; Other: Placebo; Drug: WCK 6777; Drug: Zidebactam
- Cohort 2 (Experimental): Ertapenem 2 g or placebo administered by 250 ml of intravenous infusion (IV) for 1 hour once daily for 7 days. N=8
  Interventions: Drug: Ertapenem; Other: Placebo
- Cohort 3 (Experimental): Zidebactam 2 g administered by 250 ml of intravenous infusion (IV) for 1 hour,once daily,for 7 days. N=6
  Interventions: Drug: Zidebactam
- Cohort 4 (Experimental): WCK 6777 (Ertapenem 2 g combined with Zidebactam 2 g) or placebo administered by 250 ml of intravenous infusion (IV) for 1 hour, once daily, for 7 days. N=8
  Interventions: Drug: Ertapenem; Other: Placebo; Drug: WCK 6777; Drug: Zidebactam
- Cohort 5 (Experimental): Ertapenem 3 g or placebo administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days. N=8
  Interventions: Drug: Ertapenem; Other: Placebo
- Cohort 6 (Experimental): Zidebactam 3 g administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days. N=6
  Interventions: Drug: Zidebactam
- Cohort 7 (Experimental): WCK 6777 (Ertapenem 3 g combined with Zidebactam 3 g) or placebo administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days. N=8
  Interventions: Drug: Ertapenem; Other: Placebo; Drug: WCK 6777; Drug: Zidebactam

INTERVENTIONS:
Drug: Ertapenem — A 1-beta methyl-carbapenem that is structurally related to beta-lactam antibiotics
  Arms: Cohort 1; Cohort 2; Cohort 4; Cohort 5; Cohort 7
Other: Placebo — Placebo
  Arms: Cohort 1; Cohort 2; Cohort 4; Cohort 5; Cohort 7
Drug: WCK 6777 — A combination of ertapenem (ERT) and zidebactam (ZID)
  Arms: Cohort 1; Cohort 4; Cohort 7
Drug: Zidebactam — A betaß-lactamase inhibitor and betaß-lactam enhancer from the diazabicyclooctane (DBO) class
  Arms: Cohort 1; Cohort 3; Cohort 4; Cohort 6; Cohort 7

SUMMARY:
This is a Phase 1, single center study to investigate the safety, tolerability, and pharmacokinetics (PK) of three dose-level groups of WCK 6777 (ERT and ZID combination), and two dose-level groups of ERT alone and ZID (WCK 5107) alone in 52 healthy adult male and female subjects aged 18 to 45 years old (both inclusive). Seven treatment cohorts will be evaluated in this study. WCK 6777 will be evaluated in three cohorts - Cohorts 1, 4 and 7- of 8 subjects each (6 study drug combinations and 2 placebos); ERT will be evaluated alone in two cohorts - Cohorts 2 and 5- of 8 subject each (6 ERT and 2 placebos); and ZID will be evaluated in two cohorts, Cohorts 3 and 6, of 6 subjects each (all ZID). The study will be placebo-controlled and double-blinded in all cohorts except Cohorts 3 and 6. No placebo subjects are included in standalone ZID cohorts, since adequate safety data for higher doses of ZID alone in comparison with placebo are available from completed Phase 1 studies of WCK 5107 (ZID) alone and the ZID-only arms of WCK 5222 (cefepime + ZID) studies. The primary objective is to assess the safety and tolerability of three dose-escalating regimens of WCK 6777 ( ERT and ZID combination) and two-dose escalating regimens of standalone ERT or ZID following single daily doses for 7 days in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single center study to investigate the safety, tolerability, and pharmacokinetics (PK) of three dose-level groups of WCK 6777 (ERT and ZID combination), and two dose-level groups of ERT alone and ZID (WCK 5107) alone in 52 healthy adult male and female subjects aged 18 to 45 years old (both inclusive). Seven treatment cohorts will be evaluated in this study. WCK 6777 will be evaluated in three cohorts - Cohorts 1, 4 and 7- of 8 subjects each (6 study drug combinations and 2 placebos); ERT will be evaluated alone in two cohorts - Cohorts 2 and 5- of 8 subject each (6 ERT and 2 placebos); and ZID will be evaluated in two cohorts, Cohorts 3 and 6, of 6 subjects each (all ZID). The study will be placebo-controlled and double-blinded in all cohorts except Cohorts 3 and 6. No placebo subjects are included in standalone ZID cohorts, since adequate safety data for higher doses of ZID alone in comparison with placebo are available from completed Phase 1 studies of WCK 5107 (ZID) alone and the ZID-only arms of WCK 5222 (cefepime + ZID) studies. In each cohort, either study drugs alone or their combination will be administered by a single intravenous infusion (IV) of 100 mL daily for 7 consecutive days in Cohort 1 or 250 mL daily for 7 consecutive days in Cohorts 2 to 7. For each treatment cohort, however, the dose will be progressively escalated from 1 g/daily to 2 g/daily and to 3 g/daily, and the duration of infusion time increased from 30 min to 1 h and to 2 h over the course of the study. In Cohort 1, WCK 6777 2 g (ERT 1 g/daily combined with ZID 1 g/daily) will be administered in 30 (±5) minutes (min); in Cohort 2 (ERT 2 g/daily), Cohort 3 (ZID 2 g/daily), and Cohort 4 (WCK 6777 4 g [ERT 2 g/daily combined with ZID 2 g/daily]) the study drug(s) will be administered in 60 (±10) min, and in Cohort 5 (ERT 3 g/daily), Cohort 6 (ZID 3 g daily) and Cohort 7 (WCK 6777 6 g [ERT 3 g/daily combined with ZID 3 g/daily]), the study drug(s) will be administered in 120 (±10) min. The primary objective is to assess the safety and tolerability of three dose-escalating regimens of WCK 6777 ( ERT and ZID combination) and two-dose escalating regimens of standalone ERT or ZID following single daily doses for 7 days in healthy adult subjects. The secondary objective is to characterize the PK profiles in plasma (total & free) and in urine of three dose-escalating regimens of WCK 6777 (ERT and ZID combination) and two dose-escalating regimens of standalone ERT or ZID following a single initial dose on Day 1 and after single daily doses for 7 days in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated written informed consent and agrees to comply with the study procedures and length of confinement to the research site.
2. Be able to understand and willing to comply with study procedures, restrictions, and requirements, as determined by the Site Principal Investigator (PI) or authorized clinician(s) (listed on FDA Form 1572).
3. Adults 18 to 45 years of age inclusive, including non-pregnant, non-lactating females.
4. Have suitable veins for cannulation or repeated venipuncture.
5. Be in good general health at the time of enrollment. Note 1: Determined by medical history (MH), medication use, physical examination (PE), vital signs (VS), clinical laboratory tests including estimated creatinine clearance (CLCR) > / = 80 mL/min by the Cockcroft-Gault method, and 12-lead Electrocardiogram (ECG) within reference ranges at Screening and Day-1.

   Note 2: Exceptions to Blood Pressure (BP), Heart Rate (HR) and laboratory test values being with normal ranges are:
   * Subjects with baseline HR > / = 45 to 50 Beats per Minute (bpm) may be accepted if otherwise healthy adults with known history of asymptomatic bradycardia.
   * Subjects with baseline Systolic Blood Pressure (SBP) up to 140 Millimeters of Mercury (mmHg) and Diastolic Blood Pressure (DBP) up to 90 mmHg may be accepted if otherwise healthy.
   * A laboratory value that is Grade 1 will be allowed if not considered to be clinically significant by the investigator, with the exception of Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (AP), total and direct bilirubin, Blood Urea Nitrogen (BUN), serum creatinine, Creatinine Clearance (CLcr), and urine protein.
6. Sexually active females must be of non-childbearing potential or must use a highly effective method of birth control from screening to 30 days following the last dose of study product.

   Note 1: A female is considered of childbearing potential unless post-menopausal (defined as history of > / = 1 year of spontaneous amenorrhea and a Follicle-Stimulating Hormone (FSH) level >40 IU/L), or permanently surgically sterilized.

   Note 2: Highly effective contraceptive methods include: (a) surgical sterilization methods, such as tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful tubal obliteration (e.g., Essure(R)) with documented radiological confirmation test at least 90 days after the procedure, or (b) long-acting reversible contraception, such as progestin-releasing subdermal implants, copper intrauterine devices (IUDs), levonorgestrel-releasing IUDs.

   Note 3: A subject who is not sexually active and abstains from sexual intercourse can be enrolled and abstinence documented.
7. Sexually active males must be vasectomized or agree to use barrier contraception and not donate sperm from first dose of study product until 30 days following the last dose.

   Note 1: Barrier contraception includes use of condom with spermicide. Note 2: A subject who is not sexually active and abstains from sexual intercourse can be enrolled and abstinence documented.
8. Subjects must be willing to avoid excessive physical exercise within 48 h prior to dosing until discharge from the CTU on Day 8, and 24 h before the last visit (Day 11 +3 days).
9. No history of acute febrile or infectious illness for at least 7 days prior to the administration of study drug(s).

Exclusion Criteria:

1. Known history of a clinically significant food or drug allergy/hypersensitivity including known allergy/hypersensitivity to Ertapenem (ERT), any ß-lactam drugs or other related drugs.
2. Current seasonal allergies with ongoing symptoms for more than a week prior to dosing requiring glucocorticoids and/or frequent use of antihistamines for treatment.
3. Any history of a chronic condition including renal failure that may increase risk to subject or interfere with endpoint assessment, or any unstable chronic disease.

   Note 1: Unstable chronic disease is defined by need for frequent medical interventions that lead to a change in medications and/or required hospitalization, surgery or an invasive procedure or emergency department/urgent care visit, as determined by the Site PI.

   Note 2: Any chronic disease, that has been diagnosed within 90 days of screening is excluded.
4. History of any psychiatric condition that has required hospitalization in the last 12 months or subject is considered psychologically unstable by the investigator.
5. History of any clinically significant (CS) disease or disorder, medical/surgical procedure, or trauma within 4 weeks prior to initiation of administration of study product(s).
6. History of Clostridium difficile induced diarrhea within 1 year before screening
7. Known history of past or current epilepsy or seizure disorders, excluding febrile seizures of childhood.
8. Prior exposure to Zidebactam (ZID).
9. Use of any prohibited prescription or non-prescription medication within 14 days prior to the first dose of study drug(s) as described in Section 6.6
10. Use of any investigational drug product within 30 days or 5 half-lives (whichever is longer) before investigational product administration in this study.
11. Planned participation in a clinical research study that requires treatment with a study drug, blood draws or other invasive assessments during the study period (screening until final visit).
12. Blood or plasma donation of 500 mL within 3 months or more than 100 mL within 30 days before signing informed consent or planned donation prior to completion of this trial.
13. Positive serum pregnancy test for women at screening and urine pregnancy test at check-in.
14. Positive urine alcohol test or urine drug screen test at screening or check-in (Day -1).
15. Positive test for HIV antibodies, hepatitis B-virus surface antigen (HBsAg), or anti-hepatitis C-virus antibodies (anti-HCV) at screening.
16. History of > / = 10 pack-years smoking in the 5-year period before screening, or positive urine cotinine screen at check-in.

    Note 1: Nicotine products include cigarettes, e-cigarettes, pipe, cigar, chewing tobacco, nicotine patch.

    Note 2: Positive urine cotinine at screening is allowed if negative at check-in (Day -1).
17. History of binge drinking or heavy drinking of alcohol at any time in the 6 months before study product administration.

Note 1: Binge drinking is defined as 5 or more drinks during single occasion if male, or 4 or more if female.

Note 2: Heavy drinking of alcohol is defined as consumption of more than 15 units of alcohol per week if male, or more than 8 units if female.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Inc - Kansas City, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 19APR2023 and 24OCT2023 by the clinical trials unit (CTU) utilizing the CTU subject database and IRB-approved advertisements and social media.
Groups:
- Cohort 1 - WCK 6777 2 g: WCK 6777 (Ertapenem 1 g combined with Zidebactam 1 g) administered by 100 ml of intravenous infusion (IV) for 30 (±5) minutes once daily for 7 days.
  Ertapenem: A 1-ß methyl-carbapenem that is structurally related to ß-lactam antibiotics
  Zidebactam: A ß-lactamase inhibitor and ß-lactam enhancer from the diazabicyclooctane (DBO) class
  WCK 6777: A combination of ertapenem (ERT) and zidebactam (ZID)
- Cohort 2 - ERT 2 g: Ertapenem 2 g administered by 250 ml of intravenous infusion (IV) for 1 hour once daily for 7 days.
  Ertapenem: A 1-ß methyl-carbapenem that is structurally related to ß-lactam antibiotics
- Cohort 3 - ZID 2 g: Zidebactam 2 g administered by 250 ml of intravenous infusion (IV) for 1 hour,once daily,for 7 days.
  Zidebactam: A ß-lactamase inhibitor and ß-lactam enhancer from the diazabicyclooctane (DBO) class
- Cohort 4 - WCK 6777 4 g: WCK 6777 (Ertapenem 2 g combined with Zidebactam 2 g) administered by 250 ml of intravenous infusion (IV) for 1 hour, once daily, for 7 days.
  Ertapenem: A 1-ß methyl-carbapenem that is structurally related to ß-lactam antibiotics
  Zidebactam: A ß-lactamase inhibitor and ß-lactam enhancer from the diazabicyclooctane (DBO) class
  WCK 6777: A combination of ertapenem (ERT) and zidebactam (ZID)
- Cohort 5 - ERT 3 g: Ertapenem 3 g administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
  Ertapenem: A 1-ß methyl-carbapenem that is structurally related to ß-lactam antibiotics
- Cohort 6 - ZID 3 g: Zidebactam 3 g administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
  Zidebactam: A ß-lactamase inhibitor and ß-lactam enhancer from the diazabicyclooctane (DBO) class
- Cohort 7 - WCK 6777 6 g: WCK 6777 (Ertapenem 3 g combined with Zidebactam 3 g) administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
  Ertapenem: A 1-ß methyl-carbapenem that is structurally related to ß-lactam antibiotics
  Zidebactam: A ß-lactamase inhibitor and ß-lactam enhancer from the diazabicyclooctane (DBO) class
  WCK 6777: A combination of ertapenem (ERT) and zidebactam (ZID)
- Placebo: Placebo participants from Cohorts 1,2,4,5,7. Placebo administered corresponding to method for active drug administration in each cohort.
Period: Overall Study
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Started | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Enrolled but treatment not administered | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 7 | 6 | 10 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (7.3) | 35.2 (9.2) | 32.3 (9.5) | 33.2 (7.0) | 33.6 (7.9) | 37.3 (5.6) | 29.2 (9.0) | 30.7 (6.7) | 33.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 2 | 2 | 2 | 4 | 20
  Male | 4 | 3 | 4 | 3 | 5 | 5 | 4 | 6 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 8
  Not Hispanic or Latino | 4 | 5 | 6 | 5 | 5 | 6 | 6 | 9 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 4 | 2 | 1 | 2 | 2 | 5 | 7 | 28
  White | 0 | 2 | 4 | 5 | 4 | 5 | 1 | 2 | 23
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.08 (2.93) | 28.57 (2.05) | 25.18 (3.38) | 27.63 (2.85) | 23.83 (1.62) | 27.27 (2.76) | 24.05 (4.36) | 26.87 (2.82) | 26.32 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) are defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, regardless of its causal relationship to the product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of the product, and are described as treatment-emergent AEs (TEAEs). Number of participants with a TEAE are summarized by dose group and by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - WCK 6777 2 g: WCK 6777 (Ertapenem 1 g combined with Zidebactam 1 g) administered by 100 ml of intravenous infusion (IV) for 30 (±5) minutes once daily for 7 days.
- Cohort 2 - ERT 2 g: Ertapenem 2 g administered by 250 ml of intravenous infusion (IV) for 1 hour once daily for 7 days.
- Cohort 3 - ZID 2 g: Zidebactam 2 g administered by 250 ml of intravenous infusion (IV) for 1 hour,once daily,for 7 days.
- Cohort 4 - WCK 6777 4 g: WCK 6777 (Ertapenem 2 g combined with Zidebactam 2 g) administered by 250 ml of intravenous infusion (IV) for 1 hour, once daily, for 7 days.
- Cohort 5 - ERT 3 g: Ertapenem 3 g administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
- Cohort 6 - ZID 3 g: Zidebactam 3 g administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
- Cohort 7 - WCK 6777 6 g: WCK 6777 (Ertapenem 3 g combined with Zidebactam 3 g) administered by 250 ml of intravenous infusion (IV) for 2 hours, once daily, for 7 days.
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Blood and lymphatic system disorders | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Gastrointestinal disorders | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 1
  General disorders and administration site conditions | 3 | 5 | 5 | 4 | 4 | 2 | 3 | 6
  Infections and infestations | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Investigations | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 3
  Musculoskeletal and connective tissue disorders | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system disorders | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  Renal and urinary disorders | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Treatment-Emergent Adverse Events Reported
Description: Adverse events (AEs) are defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, regardless of its causal relationship to the product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of the product, and are described as treatment-emergent AEs (TEAEs). Number of TEAEs reported are summarized by dose group and MedDRA System Organ Class (SOC)..
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Number; unit: events
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
events
  Blood and lymphatic system disorders | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Gastrointestinal disorders | 3 | 2 | 0 | 1 | 1 | 0 | 1 | 1
  General disorders and administration site conditions | 6 | 11 | 8 | 6 | 6 | 3 | 6 | 14
  Infections and infestations | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Investigations | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 3
  Musculoskeletal and connective tissue disorders | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system disorders | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  Renal and urinary disorders | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Related to Study Product
Description: Adverse events (AEs) are defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, regardless of its causal relationship to the product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of the product, and are described as treatment-emergent AEs (TEAEs). TEAEs are assessed by the investigator to determine relationship to the study drug. Number of participants with a related TEAE are summarized by dose group and by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Blood and lymphatic system disorders | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Gastrointestinal disorders | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 1
  General disorders and administration site conditions | 3 | 5 | 4 | 3 | 2 | 2 | 3 | 4
  Infections and infestations | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Investigations | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2
  Musculoskeletal and connective tissue disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  Renal and urinary disorders | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Serious Adverse Events Reported
Description: Serious AEs (SAEs) meet one or more of the following criteria: death, life-threatening AEs, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, substantial disruption of the ability to conduct normal life function, congenital anomaly/birth defect, or important medical events that may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. SAEs are listed.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Number; unit: events
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Chemistry Laboratory Toxicity Results
Description: Parameters and thresholds include alanine aminotransferase =33 (female (F) 19Y), =30 (F >19) or =47 U/L (male (M) =19Y); albumin =3.5 g/dL; alkaline phosphatase =129 (F 19Y), =126 (F =49Y), =170 (M 19Y) or =131 U/L (M =49Y); aspartate aminotransferase =33 (19Y) or =41 U/L (20-49Y); bilirubin =1.2 (19Y) or =1.3 mg/dL (>19Y); calcium =8.8 (4-19Y), =8.5 (20-49Y), =10.5 (4-19Y), =10.3 (F 20-49Y) or =10.4 mg/dL (M 20-49Y); carbon dioxide =19 or =33 mmol/L; creatinine =0.97 (F 18-29Y), =0.98 (F 30-39Y), =1.00 (F 40-49Y), =1.25 (M 18-29Y), =1.27 (M 30-39Y) or =1.30 mg/dL (M 40-49Y); direct bilirubin =0.3 mg/dL; glucose =64 or =100 mg/dL; potassium =3.7 (19Y), =3.4 (>19Y), = 5.2 (19Y) or = 5.4 mmol/L (>19Y); protein =6.2 (19Y) or =6.0 g/dL (>19Y); sodium =134 or =147 mmol/L; and urea nitrogen =21 (19Y) or =26 mg/dL (>19Y). All abnormal toxicity results are included, but Grade 1 values at screening/baseline allowed for enrollment were only considered TEAEs if they increased in severity.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Alanine aminotransferase increase | 0 | 2 | 0 | 2 | 2 | 0 | 1 | 1
  Albumin decrease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Alkaline phosphatase increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increase | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Bilirubin increase | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Calcium decrease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Calcium increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Carbon dioxide decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Carbon dioxide increase | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Creatinine increase | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Direct bilirubin increase | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose increase | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Potassium decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein decrease | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Sodium decrease | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Sodium increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea nitrogen increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Toxicity Results
Description: Parameters and thresholds include basophils =201 x106/L (>6Y); eosinophils =501 x106/L (>6Y); hemoglobin =11.4 (female (F) 18Y), =11.6 (F >18Y), =11.9 (male (M) 18Y) or =13.1 g/dL (M >18Y); leukocytes =4.4 (18Y), =3.7 (>18Y), =13.1 (18Y) or =10.9 x109/L (>18Y); lymphocytes =1199 (18Y) or =849 x106/L (>18Y); monocytes =901 (18Y) or =951 x106/L (>18Y); neutrophils =1799 (18Y) or =1499 x106/L (>18Y); and platelets <140 x109/L. All abnormal toxicity results are included, but Grade 1 values at screening/baseline allowed for enrollment were only considered TEAEs if they increased in severity.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Basophils increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin decrease | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 5
  Leukocytes decrease | 3 | 0 | 0 | 2 | 2 | 0 | 3 | 2
  Leukocytes increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils decrease | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 2
  Platelets decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Coagulation Laboratory Toxicity Results
Description: Parameters and thresholds include activated partial thromboplastin time >32 s, prothrombin intl. normalized ratio >1.1 (ratio), and prothrombin time >11.5 s. All abnormal toxicity results are included, but Grade 1 values at screening/baseline allowed for enrollment were only considered TEAEs if they increased in severity.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Activated partial thromboplastin time increase | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Prothrombin intl. normalized ratio (INR) increase | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Prothrombin time increase | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1

8. Primary Outcome: Number of Participants With Abnormal Urinalysis Laboratory Toxicity Results
Description: Parameters and thresholds include dipstick measurements of glucose =1+, leukocyte esterase =1+, occult blood =1+, protein =1+ and urinalysis with microscopy results of at least a few bacteria, red blood cells (RBC) =3 per high-powered field (HPF), and white blood cells (WBC) =6 per HPF. If dipstick results were abnormal, urinalysis with microscopy was performed. All abnormal toxicity results are included, but Grade 1 values at screening/baseline allowed for enrollment were only considered TEAEs if they increased in severity.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Glucose increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase increase | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2
  Occult blood increase | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Protein increase | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  RBC increase: number analyzed (Participants) | 2 | 4 | 1 | 2 | 0 | 1 | 1 | 3
  RBC increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WBC increase: number analyzed (Participants) | 2 | 4 | 1 | 2 | 0 | 1 | 1 | 3
  WBC increase | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1
  Bacteria increase: number analyzed (Participants) | 2 | 4 | 1 | 2 | 0 | 1 | 1 | 3
  Bacteria increase | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3

9. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Toxicity Results
Description: The only ECG parameters graded were PR interval with a threshold of =211 msec and QTcF interval with a threshold of =471 msec (female) or =451 msec (male) or an increase of =30 msec above baseline. ECG values after dosing were considered as TEAEs if they met toxicity grading criteria.
Time Frame: Day 8 and Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  PR interval | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Vital Signs (VS)
Description: VS parameters and thresholds include diastolic blood pressure =90 mmHg, oral temperature =37.3 °C, pulse =49 or =101 beats/min, respiratory rate =21 breaths/min, and systolic blood pressure =88 or =131 mmHg. VS could be repeated up to twice more at rest and within at least 5 minutes of each other. The following rules were used to determine which vital sign measurement to use for analysis if repeat measurements occurred: 1. If the first replicate was normal, it was used. 2. If the first and second replicates were both abnormal, the replicate with the higher severity was used. 3. If the first replicate was abnormal, the second replicate was normal, and the third replicate was not performed, the first replicate was used. 4. If the first replicate was abnormal and the second and third replicates were normal, the second replicate was used. 5. If the first and third replicates were abnormal and the second replicate was normal, the abnormal replicate with the higher severity was used.
Time Frame: Day 1 through Day 11
Population: Safety Population: All participants that received any amount of study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Diastolic blood pressure increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Oral temperature increase | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Pulse decrease | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Pulse increase | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Respiratory rate increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure increase | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1

11. Secondary Outcome: Maximum Observed Concentration (Cmax) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the Cmax (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group.
Time Frame: =0.5 h prior to dosing and 0.25 h (WCK 6777 2g group only), 0.5 h (WCK 6777 2g, ERT 2g, ZID 2g, and WCK 6777 4g groups only), 1 h, 2 h, 3 h, 4 h, 8 h, 12 h, 18 h, and 24 h post-start of Dose 1 (Day 1) infusion
Population: PK Analysis Subset Population: all participants who received the intended dose of study drug(s) on the given day(s) of analysis, have at least one quantifiable post-dosing plasma drug concentration measured, and have sufficient data that permit estimation of PK parameters. Any participant with at least one estimable PK parameter is included in this subset.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 196.66 (14) | 303.43 (9) |  | 354.41 (8) | 378.71 (10) |  | 391.87 (13)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 16.60 (17) | 34.00 (17) |  | 42.10 (22) | 58.45 (17) |  | 59.42 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 69.67 (15) |  | 120.41 (22) | 133.51 (16) |  | 111.71 (10) | 128.42 (11)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 64.35 (20) |  | 105.42 (16) | 98.41 (55) |  | 108.79 (11) | 124.99 (10)

12. Secondary Outcome: Minimum Observed Concentration (Cmin) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the Cmin (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 2.15 (50) | 2.61 (107) |  | 3.10 (60) | 7.32 (14) |  | 5.91 (33)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.10 (40) | 0.16 (42) |  | 0.14 (67) | 0.36 (24) |  | 0.28 (35)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.09 (37) |  | 0.11 (72) | 0.10 (44) |  | 0.13 (28) | 0.15 (30)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.09 (22) |  | 0.07 (36) | 0.10 (39) |  | 0.14 (26) | 0.14 (34)

13. Secondary Outcome: Predicted Concentration at the End of the Dosing Interval (Ctau) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the Ctau (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group. Ctau is estimated using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 2.02 (50) | 2.29 (112) |  | 2.83 (61) | 6.83 (16) |  | 5.44 (34)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.08 (39) | 0.10 (102) |  | 0.13 (67) | 0.31 (23) |  | 0.27 (38)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.02 (101) |  | 0.06 (69) | 0.05 (87) |  | 0.11 (33) | 0.13 (31)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.04 (102) |  | 0.06 (49) | 0.05 (96) |  | 0.11 (34) | 0.12 (34)

14. Secondary Outcome: Dose-Normalized Maximum Observed Concentration (Cmax/Dose) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the dose-normalized Cmax ((µg/mL)/mg) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (µg/mL)/mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
(µg/mL)/mg
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 0.20 (14) | 0.15 (9) |  | 0.18 (8) | 0.13 (10) |  | 0.13 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.02 (17) | 0.02 (17) |  | 0.02 (22) | 0.02 (17) |  | 0.02 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.07 (15) |  | 0.06 (22) | 0.07 (16) |  | 0.04 (10) | 0.04 (11)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.06 (20) |  | 0.05 (16) | 0.05 (55) |  | 0.04 (11) | 0.04 (10)

15. Secondary Outcome: Time of Maximum Concentration (Tmax) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Median and minimum/maximum of the Tmax (h) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 0.50 [0.50 to 0.50] | 1.00 [1.00 to 1.07] |  | 1.00 [1.00 to 1.00] | 2.02 [2.00 to 2.03] |  | 2.03 [2.02 to 2.03]
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.50 [0.50 to 0.50] | 1.00 [1.00 to 1.07] |  | 1.00 [1.00 to 1.00] | 2.02 [2.02 to 2.03] |  | 2.03 [2.02 to 2.03]
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.50 [0.50 to 0.50] |  | 1.03 [1.02 to 1.03] | 1.00 [1.00 to 1.00] |  | 2.02 [1.03 to 2.02] | 2.03 [2.02 to 2.03]
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.50 [0.50 to 0.50] |  | 1.03 [1.02 to 1.03] | 1.00 [1.00 to 2.00] |  | 2.02 [1.03 to 2.02] | 2.03 [2.02 to 2.03]

16. Secondary Outcome: Time of Minimum Concentration (Tmin) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Median and minimum/maximum of the Tmin (h) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 23.60 [23.60 to 23.70] | 23.65 [23.60 to 23.70] |  | 23.60 [23.60 to 23.60] | 23.60 [23.40 to 23.60] |  | 23.60 [23.60 to 23.70]
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 23.60 [18.00 to 23.60] | 23.60 [18.00 to 23.70] |  | 23.60 [23.60 to 23.60] | 23.60 [23.40 to 23.60] |  | 23.60 [23.60 to 23.70]
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 18.00 [18.00 to 23.60] |  | 23.60 [18.00 to 23.70] | 23.60 [18.00 to 23.60] |  | 23.60 [23.60 to 23.60] | 23.60 [23.60 to 23.70]
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 23.60 [18.00 to 23.70] |  | 23.60 [23.60 to 23.70] | 23.60 [18.00 to 23.60] |  | 23.60 [23.60 to 23.60] | 23.60 [23.60 to 23.70]

17. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing to the Predicted Time the Concentration Reaches the Lower Limit of Quantification (AUC(0-t)) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total area under the concentration-time curve from dosing (time 0 h) extrapolated to the time the concentration is predicted to reach the lower limit of quantification (LLOQ), AUC(0-t) (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 723.48 (9) | 1241.47 (18) |  | 1377.99 (14) | 2148.23 (11) |  | 2024.46 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 39.92 (7) | 83.95 (19) |  | 102.81 (24) | 187.42 (15) |  | 190.43 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 140.00 (8) |  | 302.40 (18) | 320.50 (20) |  | 379.92 (9) | 442.32 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 125.17 (8) |  | 257.74 (15) | 247.40 (42) |  | 379.75 (11) | 427.31 (16)

18. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing to Time of the Last Measured Concentration (AUC(0-last)) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total area under the concentration-time curve from dosing (time 0 h) to the time of last measured concentration, AUC(0-last) (µg*h/mL),parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 728.18 (9) | 1247.86 (18) |  | 1384.69 (14) | 2153.20 (11) |  | 2027.57 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 41.04 (7) | 85.03 (19) |  | 103.94 (23) | 188.66 (15) |  | 191.81 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 141.17 (8) |  | 303.42 (18) | 321.35 (20) |  | 381.44 (9) | 443.70 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 126.34 (8) |  | 259.11 (15) | 248.60 (42) |  | 380.91 (11) | 428.67 (16)

19. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing Taken to the Limit as the End Time Becomes Arbitrarily Large (AUC(0-inf)) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total area under the concentration-time curve from dosing (time 0 h) taken to the limit as the end time becomes arbitrarily large, AUC(0-inf) (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 742.95 (10) | 1265.39 (19) |  | 1404.86 (15) | 2199.93 (11) |  | 2065.37 (11)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 41.65 (7) | 85.93 (19) |  | 104.94 (24) | 190.81 (15) |  | 193.61 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 141.33 (8) |  | 303.92 (18) | 322.04 (20) |  | 381.76 (9) | 444.34 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 126.50 (8) |  | 259.27 (15) | 249.11 (41) |  | 381.44 (11) | 429.33 (16)

20. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing Extrapolated to 24 Hours After Dosing (AUC(0-24)) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total area under the concentration-time curve from dosing (time 0 h) extrapolated to 24 h after dosing, AUC(0-24) (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 728.97 (9) | 1249.60 (18) |  | 1386.28 (14) | 2156.38 (11) |  | 2029.12 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 41.19 (7) | 85.25 (19) |  | 103.96 (23) | 188.86 (15) |  | 192.13 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 141.17 (8) |  | 303.60 (18) | 321.76 (20) |  | 381.59 (9) | 443.70 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 126.34 (8) |  | 259.11 (15) | 248.60 (42) |  | 380.91 (11) | 428.67 (16)

21. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing to the End of the Dosing Interval (AUC(0-tau)) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total area under the concentration-time curve from dosing (time 0 h) to the end of the dosing interval (24 h post-infusion), AUC(0-tau) (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 728.97 (9) | 1249.60 (18) |  | 1386.28 (14) | 2156.38 (11) |  | 2029.12 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 41.19 (7) | 85.25 (19) |  | 103.96 (23) | 188.86 (15) |  | 192.13 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 141.17 (8) |  | 303.60 (18) | 321.76 (20) |  | 381.59 (9) | 443.70 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 126.34 (8) |  | 259.11 (15) | 248.60 (42) |  | 380.91 (11) | 428.67 (16)

22. Secondary Outcome: Dose-Normalized Area Under the Concentration-Time Curve From Dosing to the End of the Dosing Interval (AUC(0-tau)/Dose) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the dose-normalized total area under the concentration-time curve from dosing (time 0 h) to the end of the dosing interval (24 h post-infusion), AUC(0-tau)/Dose ((µg*h/mL)/mg), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (µg*h/mL)/mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
(µg*h/mL)/mg
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 0.73 (9) | 0.62 (18) |  | 0.69 (15) | 0.72 (11) |  | 0.68 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.04 (7) | 0.04 (19) |  | 0.05 (24) | 0.06 (15) |  | 0.06 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.14 (8) |  | 0.15 (18) | 0.16 (20) |  | 0.13 (9) | 0.15 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.13 (8) |  | 0.13 (15) | 0.12 (41) |  | 0.13 (11) | 0.14 (16)

23. Secondary Outcome: Terminal Elimination Half-Life (t1/2) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the terminal elimination half-life, t1/2 (h), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 4.34 (12) | 3.76 (22) |  | 3.92 (14) | 4.20 (4) |  | 4.20 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 4.09 (11) | 3.83 (21) |  | 3.86 (15) | 3.96 (12) |  | 3.87 (10)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 2.35 (15) |  | 2.60 (14) | 2.57 (12) |  | 2.61 (9) | 2.71 (6)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 2.75 (18) |  | 2.81 (14) | 2.63 (15) |  | 2.69 (9) | 2.71 (5)

24. Secondary Outcome: Total Clearance (CLT) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total clearance, CLT (L/h), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 1.34 (10) | 1.58 (19) |  | 1.42 (15) | 1.37 (11) |  | 1.45 (11)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 23.99 (7) | 23.28 (19) |  | 19.06 (24) | 15.70 (15) |  | 15.50 (14)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 7.07 (8) |  | 6.58 (18) | 6.21 (20) |  | 7.86 (9) | 6.75 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 7.91 (8) |  | 7.71 (15) | 8.03 (41) |  | 7.86 (11) | 6.99 (16)

25. Secondary Outcome: First-Order Terminal Phase Elimination Rate Constant (Ke) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the first-order terminal phase elimination rate constant, Ke (1/h), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
1/h
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 0.16 (12) | 0.18 (22) |  | 0.18 (14) | 0.17 (4) |  | 0.17 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.17 (11) | 0.18 (21) |  | 0.18 (15) | 0.18 (12) |  | 0.18 (10)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.30 (15) |  | 0.27 (14) | 0.27 (12) |  | 0.27 (9) | 0.26 (6)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.25 (18) |  | 0.25 (14) | 0.26 (14) |  | 0.26 (9) | 0.26 (5)

26. Secondary Outcome: Apparent Volume of Distribution (Vd) for Dose 1 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the apparent volume of distribution, Vd (L), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 1 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Total ERT | 8.43 (7) | 8.57 (9) |  | 8.04 (12) | 8.28 (10) |  | 8.81 (13)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 141.43 (11) | 128.25 (12) |  | 106.20 (23) | 89.98 (20) |  | 86.55 (16)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 23.97 (14) |  | 24.67 (28) | 23.05 (22) |  | 29.56 (10) | 26.43 (16)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 31.37 (12) |  | 31.18 (23) | 30.42 (40) |  | 30.52 (9) | 27.28 (17)

27. Secondary Outcome: Maximum Observed Concentration at Steady State (Cmax,ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the Cmax,ss (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group. These estimates assume steady state has been achieved.
Time Frame: =0.5 h prior to the start of Dose 7 (Day 7) dosing and 0.25 h (WCK 6777 2g group only), 0.5 h (WCK 6777 2g, ERT 2g, ZID 2g, and WCK 6777 4g groups only), 1 h, 2 h, 3 h, 4 h, 8 h, 12 h, 18 h, and 24 h post-start of Dose 7 infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 181.90 (11) | 341.92 (10) |  | 344.89 (10) | 387.57 (9) |  | 343.24 (13)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Free ERT | 15.41 (24) | 38.18 (13) |  | 36.09 (23) | 57.65 (28) |  | 50.36 (28)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 63.87 (17) |  | 115.71 (16) | 130.69 (18) |  | 109.41 (7) | 113.79 (16)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 57.89 (23) |  | 103.12 (18) | 83.36 (57) |  | 111.59 (7) | 111.81 (16)

28. Secondary Outcome: Minimum Observed Concentration at Steady State (Cmin,ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the Cmin,ss (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group. These estimates assume steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 1.75 (30) | 1.81 (114) |  | 1.74 (75) | 4.93 (2) |  | 3.49 (65)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.10 (28) | 0.12 (35) |  | 0.12 (60) | 0.23 (31) |  | 0.15 (59)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.13 (49) |  | 0.12 (68) | 0.10 (46) |  | 0.13 (27) | 0.12 (36)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.12 (66) |  | 0.10 (38) | 0.17 (864) |  | 0.14 (23) | 0.11 (34)

29. Secondary Outcome: Dose-Normalized Maximum Observed Concentration at Steady State (Cmax,ss/Dose) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the dose-normalized Cmax,ss ((µg/mL)/mg) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group. This estimate assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (µg/mL)/mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
(µg/mL)/mg
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.18 (11) | 0.17 (10) |  | 0.17 (10) | 0.13 (9) |  | 0.11 (13)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.02 (24) | 0.02 (13) |  | 0.02 (23) | 0.02 (28) |  | 0.02 (28)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.06 (17) |  | 0.06 (16) | 0.07 (18) |  | 0.04 (7) | 0.04 (16)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.06 (23) |  | 0.05 (18) | 0.04 (56) |  | 0.04 (7) | 0.04 (15)

30. Secondary Outcome: Average Concentration Over the Dose 7 Dosing Interval (Cavg) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the average concentration over the Dose 7 dosing interval, Cavg (µg/mL) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). Cavg is calculated as AUC(0-tau,ss)/tau. These estimates assume steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 29.99 (9) | 51.20 (13) |  | 51.40 (16) | 80.91 (6) |  | 71.98 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 1.64 (6) | 3.51 (18) |  | 3.77 (16) | 7.01 (23) |  | 6.29 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 5.56 (8) |  | 11.94 (20) | 12.83 (19) |  | 16.05 (7) | 16.52 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 5.03 (8) |  | 10.48 (20) | 9.77 (30) |  | 16.32 (8) | 15.83 (14)

31. Secondary Outcome: Predicted Concentration at the End of the Dosing Interval at Steady State (Ctau,ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the predicted concentration at the end of the dosing interval at steady state, Ctau,ss (µg/mL), parameters estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). These estimates assume steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
µg/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 1.75 (30) | 1.85 (111) |  | 1.74 (75) | 4.93 (2) |  | 3.50 (64)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.06 (53) | 0.07 (128) |  | 0.07 (88) | 0.23 (31) |  | 0.15 (58)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.02 (68) |  | 0.06 (89) | 0.05 (176) |  | 0.13 (28) | 0.12 (35)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.06 (169) |  | 0.07 (90) | 0.11 (2318) |  | 0.14 (23) | 0.11 (34)

32. Secondary Outcome: Time of Maximum Concentration at Steady State (Tmax,ss) for Dose 7 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Median and minimum/maximum of the Tmax,ss (h) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group. The estimate for Tmax,ss assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.52 [0.50 to 0.60] | 1.00 [1.00 to 1.00] |  | 1.02 [1.00 to 1.02] | 2.02 [2.02 to 2.02] |  | 2.07 [2.02 to 2.23]
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.52 [0.25 to 0.60] | 1.00 [1.00 to 1.00] |  | 1.02 [0.50 to 1.02] | 2.02 [2.02 to 2.02] |  | 2.07 [2.02 to 2.23]
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.52 [0.25 to 0.60] |  | 1.00 [1.00 to 1.00] | 1.02 [1.00 to 1.02] |  | 2.02 [2.02 to 2.07] | 2.07 [2.02 to 2.23]
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.52 [0.25 to 0.60] |  | 1.00 [1.00 to 1.00] | 1.02 [1.00 to 2.00] |  | 2.02 [2.02 to 2.07] | 2.07 [2.02 to 2.23]

33. Secondary Outcome: Time of Minimum Concentration (Tmin) for Dose 7 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Median and minimum/maximum of the Tmin (h) parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 24.00 [24.00 to 24.00] | 24.05 [24.00 to 24.30] |  | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00] |  | 24.00 [24.00 to 24.10]
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 24.00 [18.00 to 24.00] | 24.00 [18.00 to 24.10] |  | 24.00 [18.00 to 24.00] | 24.00 [24.00 to 24.00] |  | 24.00 [24.00 to 24.10]
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 18.00 [18.00 to 24.00] |  | 24.00 [18.00 to 24.00] | 24.00 [18.00 to 24.00] |  | 24.00 [24.00 to 24.10] | 24.00 [24.00 to 24.10]
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 24.00 [18.00 to 24.00] |  | 24.00 [18.10 to 24.00] | 24.00 [18.00 to 24.00] |  | 24.00 [24.00 to 24.10] | 24.00 [24.00 to 24.10]

34. Secondary Outcome: Area Under the Concentration-Time Curve From Dose 7 Dosing Extrapolated to 24 Hours After Dosing at Steady State (AUC(0-24),ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the area under the concentration-time curve from dosing (time 0 h) extrapolated to 24 h after dosing at steady state, AUC(0-24),ss (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). This estimate assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 719.86 (9) | 1228.88 (14) |  | 1233.66 (16) | 1940.84 (6) |  | 1726.43 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 39.48 (6) | 84.22 (18) |  | 90.51 (16) | 168.05 (23) |  | 150.93 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 133.35 (8) |  | 286.34 (20) | 308.35 (19) |  | 384.53 (7) | 396.60 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 120.70 (8) |  | 251.56 (20) | 234.14 (30) |  | 392.09 (8) | 380.11 (14)

35. Secondary Outcome: Area Under the Concentration-Time Curve From Dose 7 Dosing to the End of the Dosing Interval at Steady State (AUC(0-tau),ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the area under the concentration-time curve from dosing (time 0 h) to the end of the dosing interval (24 h post-infusion) at steady state, AUC(0-tau),ss (µg*h/mL), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). This estimate assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
µg*h/mL
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 719.86 (9) | 1228.88 (14) |  | 1233.66 (16) | 1940.84 (6) |  | 1726.43 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 39.48 (6) | 84.22 (18) |  | 90.51 (16) | 168.05 (23) |  | 150.93 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 133.35 (8) |  | 286.34 (20) | 308.35 (19) |  | 384.53 (7) | 396.60 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 120.70 (8) |  | 251.56 (20) | 234.14 (30) |  | 392.09 (8) | 380.11 (14)

36. Secondary Outcome: Dose-Normalized Area Under the Concentration-Time Curve From Dose 7 Dosing to the End of the Dosing Interval at Steady State (AUC(0-tau),ss/Dose) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the dose-normalized total area under the concentration-time curve from dosing (time 0 h) to the end of the dosing interval (24 h post-infusion) at steady state, AUC(0-tau),ss/Dose ((µg*h/mL)/mg), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). This estimate assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (µg*h/mL)/mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
(µg*h/mL)/mg
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.72 (9) | 0.61 (13) |  | 0.62 (16) | 0.65 (6) |  | 0.58 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.04 (6) | 0.04 (18) |  | 0.05 (16) | 0.06 (23) |  | 0.05 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.13 (8) |  | 0.14 (20) | 0.15 (19) |  | 0.13 (7) | 0.13 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.12 (8) |  | 0.13 (20) | 0.12 (30) |  | 0.13 (8) | 0.13 (14)

37. Secondary Outcome: Terminal Elimination Half-Life (t1/2) for Dose 7 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the terminal elimination half-life, t1/2 (h), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
hours
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 3.91 (8) | 3.64 (19) |  | 3.67 (21) | 4.14 (4) |  | 3.86 (18)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 3.89 (19) | 3.45 (19) |  | 3.38 (19) | 3.77 (10) |  | 3.76 (17)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 2.32 (15) |  | 2.64 (12) | 2.47 (24) |  | 2.69 (3) | 2.65 (10)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 2.55 (11) |  | 2.78 (15) | 3.13 (55) |  | 2.65 (7) | 2.70 (8)

38. Secondary Outcome: Total Clearance (CLT) for Dose 7 of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the total clearance, CLT (L/h), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration).
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
L/h
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 1.39 (9) | 1.63 (13) |  | 1.62 (16) | 1.55 (7) |  | 1.74 (14)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 25.35 (6) | 23.75 (18) |  | 22.09 (16) | 17.83 (23) |  | 19.86 (19)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 7.50 (8) |  | 6.98 (20) | 6.49 (19) |  | 7.80 (7) | 7.56 (14)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 8.28 (8) |  | 7.96 (20) | 8.54 (30) |  | 7.65 (8) | 7.89 (14)

39. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vd,ss) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the apparent volume of distribution at steady state, Vd,ss (L), parameter estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h period following Dose 7 by dose group using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). This estimate assumes steady state has been achieved.
Time Frame: as for outcome 27
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
liters
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 6.86 (5) | 6.73 (11) |  | 6.51 (11) | 7.17 (9) |  | 7.58 (10)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 105.98 (14) | 72.51 (16) |  | 69.65 (13) | 56.84 (30) |  | 61.59 (29)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 18.04 (14) |  | 16.57 (18) | 13.88 (21) |  | 20.33 (7) | 19.35 (13)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 21.86 (10) |  | 18.79 (14) | 30.21 (197) |  | 20.17 (6) | 19.69 (13)

40. Secondary Outcome: Linearity Index of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the linearity index (ratio) for the total ERT, free ERT, total ZID, and free ZID plasma concentration-time data by dose group. The linearity index is a measure of how linear the relationship is between increase in administered dose and increase in exposure. The linearity index is estimated as AUC(0-tau),ss (Dose 7)/AUC(0-inf) (Dose 1), where the areas under the concentration-time curves from Dose 7 to the end of the dosing interval at steady state and from Dose 1 taken to the limit as the end time becomes arbitrarily large, AUC(0-tau),ss and AUC(0-inf) respectively, are calculated using Phoenix WinNonlin Non-compartmental Analysis with Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). The AUC(0-tau),ss estimate assumes steady state was reached.
Time Frame: =0.5 h prior to the start of and 0.25 h (WCK 6777 2g group only), 0.5 h (WCK 6777 2g, ERT 2g, ZID 2g, and WCK 6777 4g groups only), 1 h, 2 h, 3 h, 4 h, 8 h, 12 h, 18 h, and 24 h post-start of Dose 1 (Day 1) and Dose 7 (Day 7) infusions
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
ratio
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.97 (4) | 0.97 (7) |  | 0.88 (11) | 0.89 (6) |  | 0.84 (9)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.95 (4) | 0.98 (4) |  | 0.86 (18) | 0.88 (9) |  | 0.78 (17)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.94 (4) |  | 0.94 (13) | 0.96 (5) |  | 1.01 (8) | 0.89 (11)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.95 (5) |  | 0.97 (13) | 0.94 (26) |  | 1.03 (7) | 0.89 (13)

41. Secondary Outcome: The Accumulation Ratio of the Area Under the Concentration-Time Curve (RAUC) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the accumulation ratio of the AUC, RAUC (ratio), parameter for the total ERT, free ERT, total ZID, and free ZID plasma concentration-time data by dose group. RAUC is estimated as AUC(0-tau),ss (Dose 7)/AUC(0-24) (Dose 1), where the areas under the concentration-time curves from Dose 7 to the end of the dosing interval at steady state and from Dose 1 extrapolated to 24 h after Dose 1, AUC(0-tau),ss and AUC(0-24) respectively, are calculated using Phoenix WinNonlin Non-compartmental Analysis with the Ke (first-order terminal phase elimination rate constant) acceptance criteria: Rsq_adjusted (adjusted R-squared) = 0.90 and includes at least 3 timepoints after Tmax (time of maximum concentration). The AUC(0-tau),ss estimate assumes steady state was reached.
Time Frame: as for outcome 40
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
ratio
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.99 (5) | 0.98 (7) |  | 0.89 (11) | 0.91 (6) |  | 0.85 (9)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.96 (4) | 0.99 (3) |  | 0.87 (18) | 0.89 (9) |  | 0.79 (17)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.94 (4) |  | 0.94 (13) | 0.96 (5) |  | 1.01 (8) | 0.89 (11)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.96 (5) |  | 0.97 (13) | 0.94 (26) |  | 1.03 (7) | 0.89 (13)

42. Secondary Outcome: The Accumulation Ratio of the Maximum Observed Concentration (RCmax) of Total ERT, Free ERT, Total ZID, and Free ZID in Plasma
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of the accumulation ratio of the Cmax, RCmax (ratio), parameter for the total ERT, free ERT, total ZID, and free ZID plasma concentration-time data by dose group. RCmax is estimated as Cmax (Dose 7)/Cmax (Dose 1), where the Cmax parameters are estimated from the total ERT, free ERT, total ZID, or free ZID plasma concentration-time data over the 24-h periods following Dose 1 and Dose 7, respectively.
Time Frame: as for outcome 40
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
ratio
  Total ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Total ERT | 0.92 (17) | 1.13 (14) |  | 0.97 (7) | 1.01 (8) |  | 0.88 (8)
  Free ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 5 | 0 | 6
  Free ERT | 0.93 (11) | 1.12 (7) |  | 0.86 (37) | 0.99 (12) |  | 0.85 (28)
  Total ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Total ZID | 0.92 (15) |  | 0.96 (11) | 0.98 (12) |  | 0.98 (13) | 0.89 (17)
  Free ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Free ZID | 0.90 (15) |  | 0.98 (11) | 0.85 (40) |  | 1.03 (10) | 0.89 (13)

43. Secondary Outcome: Amounts of Unchanged ERT and Unchanged ZID Excreted in Urine (Ae,Urine) During Each Nominal Time Collection Interval Following Dose 1
Description: Mean and minimum/maximum of the amount of unchanged ERT and the amount of unchanged ZID excreted in urine, Ae,urine (mg), during 0-4 h, 4-8 h, 8-12 h, and 12-24 h following Dose 1 by dose group. Ae,urine parameters are calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 1 (Day 1) infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Unchanged ERT - 0-4 h: number analyzed (Participants) | 6 | 5 | 0 | 6 | 5 | 0 | 6
  Unchanged ERT - 0-4 h | 339.62 [97.70 to 605.00] | 748.60 [573.00 to 995.00] |  | 794.50 [414.00 to 1620.00] | 768.60 [451.00 to 1090.00] |  | 670.13 [87.80 to 1630.00]
  Unchanged ERT - 4-8 h: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT - 4-8 h | 159.23 [74.20 to 268.00] | 275.67 [105.00 to 414.00] |  | 202.67 [163.00 to 272.00] | 713.50 [393.00 to 1850.00] |  | 605.83 [246.00 to 1390.00]
  Unchanged ERT - 8-12 h: number analyzed (Participants) | 5 | 5 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT - 8-12 h | 64.30 [19.80 to 83.80] | 122.38 [58.80 to 204.00] |  | 128.93 [77.50 to 202.00] | 173.50 [128.00 to 227.00] |  | 192.00 [112.00 to 305.00]
  Unchanged ERT - 12-24 h: number analyzed (Participants) | 5 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT - 12-24 h | 49.80 [25.60 to 66.50] | 84.22 [49.90 to 150.00] |  | 54.38 [19.20 to 106.00] | 149.15 [84.50 to 235.00] |  | 106.95 [58.50 to 158.00]
  Unchanged ZID - 0-4 h: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 0-4 h | 544.83 [259.00 to 816.00] |  | 1336.67 [1060.00 to 1620.00] | 1475.00 [1080.00 to 2040.00] |  | 1838.33 [1270.00 to 2110.00] | 1366.50 [248.00 to 2080.00]
  Unchanged ZID - 4-8 h: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 4-8 h | 150.55 [62.60 to 277.00] |  | 360.00 [250.00 to 552.00] | 259.00 [149.00 to 314.00] |  | 631.67 [324.00 to 810.00] | 1006.00 [528.00 to 2600.00]
  Unchanged ZID - 8-12 h: number analyzed (Participants) | 5 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 8-12 h | 33.28 [6.88 to 51.30] |  | 80.35 [56.90 to 162.00] | 83.72 [38.20 to 123.00] |  | 143.50 [104.00 to 254.00] | 167.67 [127.00 to 216.00]
  Unchanged ZID - 12-24 h: number analyzed (Participants) | 3 | 0 | 5 | 4 | 0 | 6 | 6
  Unchanged ZID - 12-24 h | 19.93 [13.30 to 24.30] |  | 27.02 [15.10 to 54.10] | 25.53 [18.00 to 37.00] |  | 75.35 [37.60 to 110.00] | 75.83 [21.50 to 176.00]

44. Secondary Outcome: Cumulative Amounts of Unchanged ERT and Unchanged ZID Excreted in Urine From Zero (Predose) to 24 h Following Dose 1 (Ae,Urine(0-24))
Description: Mean and minimum/maximum of the cumulative amount of unchanged ERT and the cumulative amount of unchanged ZID excreted in urine from zero (predose) to 24 h following Dose 1, Ae,urine(0-24) (mg), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 1 (Day 1) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 1 infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT | 594.00 [204.00 to 856.00] | 1085.67 [321.00 to 1490.00] |  | 1181.83 [711.00 to 2190.00] | 1676.67 [1200.00 to 2160.00] |  | 1572.17 [843.00 to 2400.00]
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID | 733.17 [370.00 to 922.00] |  | 1798.33 [1470.00 to 1960.00] | 1836.67 [1420.00 to 2420.00] |  | 2688.33 [1820.00 to 3090.00] | 2620.00 [1040.00 to 3180.00]

45. Secondary Outcome: Fractions (%) of ERT and ZID Excreted Unchanged in Urine (fe,Urine) During Each Nominal Time Collection Interval Following Dose 1
Description: Mean and minimum/maximum of the fraction of ERT and the fraction of ZID excreted unchanged in urine, fe,urine (%), during 0-4 h, 4-8 h, 8-12 h, and 12-24 h following Dose 1 by dose group. These fe,urine parameters are calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 1 (Day 1) infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: % of dose excreted unchanged
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
% of dose excreted unchanged
  Unchanged ERT- 0-4 h: number analyzed (Participants) | 6 | 5 | 0 | 6 | 5 | 0 | 6
  Unchanged ERT- 0-4 h | 33.96 [9.77 to 60.50] | 37.46 [28.70 to 49.80] |  | 39.75 [20.70 to 81.20] | 25.60 [15.00 to 36.20] |  | 22.33 [2.93 to 54.30]
  Unchanged ERT- 4-8 h: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT- 4-8 h | 15.92 [7.42 to 26.80] | 13.78 [5.27 to 20.70] |  | 10.14 [8.14 to 13.60] | 23.77 [13.10 to 61.60] |  | 20.16 [8.18 to 46.20]
  Unchanged ERT- 8-12 h: number analyzed (Participants) | 5 | 5 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT- 8-12 h | 6.43 [1.98 to 8.38] | 6.12 [2.94 to 10.20] |  | 6.45 [3.88 to 10.10] | 5.79 [4.28 to 7.57] |  | 6.41 [3.74 to 10.20]
  Unchanged ERT- 12-24 h: number analyzed (Participants) | 5 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT- 12-24 h | 4.98 [2.56 to 6.65] | 4.21 [2.49 to 7.48] |  | 2.72 [0.96 to 5.32] | 4.97 [2.82 to 7.83] |  | 3.57 [1.95 to 5.28]
  Unchanged ZID - 0-4 h: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 0-4 h | 54.48 [25.90 to 81.60] |  | 66.70 [52.80 to 81.00] | 73.75 [54.20 to 102.00] |  | 61.25 [42.20 to 70.40] | 45.58 [8.26 to 69.40]
  Unchanged ZID - 4-8 h: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 4-8 h | 15.06 [6.26 to 27.70] |  | 17.98 [12.50 to 27.60] | 12.96 [7.45 to 15.70] |  | 21.07 [10.80 to 27.00] | 33.55 [17.60 to 86.80]
  Unchanged ZID - 8-12 h: number analyzed (Participants) | 5 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 8-12 h | 3.33 [0.69 to 5.13] |  | 4.02 [2.84 to 8.11] | 4.18 [1.91 to 6.13] |  | 4.77 [3.45 to 8.46] | 5.60 [4.22 to 7.22]
  Unchanged ZID - 12-24 h: number analyzed (Participants) | 3 | 0 | 5 | 4 | 0 | 6 | 6
  Unchanged ZID - 12-24 h | 1.99 [1.33 to 2.43] |  | 1.35 [0.76 to 2.70] | 1.27 [0.90 to 1.85] |  | 2.51 [1.25 to 3.65] | 2.53 [0.72 to 5.86]

46. Secondary Outcome: Fractions (%) of ERT and ZID Excreted Unchanged in Urine From Zero (Predose) to 24 h Following Dose 1 (fe,Urine(0-24))
Description: Mean and minimum/maximum of the fraction of ERT and the fraction of ZID excreted unchanged in urine from zero (predose) to 24 h following Dose 1, fe,urine(0-24) (%), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 1 (Day 1) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 1 infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: % of dose excreted unchanged
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
% of dose excreted unchanged
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT | 59.40 [20.40 to 85.60] | 54.32 [16.10 to 74.70] |  | 58.98 [35.50 to 109.00] | 55.85 [40.10 to 71.80] |  | 52.43 [28.10 to 79.90]
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID | 73.32 [37.00 to 92.20] |  | 89.82 [73.30 to 97.90] | 91.75 [70.90 to 121.00] |  | 89.58 [60.60 to 103.00] | 87.32 [34.50 to 106.00]

47. Secondary Outcome: Renal Clearance of ERT and ZID From Dosing Until the Last Collected Concentration for Dose 1 (CLR(0-24))
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of renal clearance of ERT and ZID from dosing until the last collected concentration for Dose 1 (24 h postdose), CLR(0-24) (mL/h ), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 1 (Day 1) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 1 infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 6 | 6 | 0 | 6
  Unchanged ERT | 0.75 (61) | 0.78 (57) |  | 0.79 (41) | 0.76 (19) |  | 0.73 (42)
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID | 4.98 (39) |  | 5.88 (15) | 5.63 (36) |  | 6.95 (25) | 5.55 (31)

48. Secondary Outcome: Amounts of Unchanged ERT and Unchanged ZID Excreted in Urine (Ae,Urine) During Each Nominal Time Collection Interval Following Dose 7
Description: Mean and minimum/maximum of the amount of unchanged ERT and the amount of unchanged ZID excreted in urine, Ae,urine (mg), during 0-4 h, 4-8 h, 8-12 h, and 12-24 h following Dose 7 by dose group. Ae,urine parameters are calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 7 (Day 7) infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
mg
  Unchanged ERT - 0-4 h: number analyzed (Participants) | 6 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 0-4 h | 357.83 [208.00 to 525.00] | 702.30 [39.50 to 1270.00] |  | 777.80 [433.00 to 1490.00] | 1010.40 [655.00 to 1530.00] |  | 998.17 [467.00 to 1670.00]
  Unchanged ERT - 4-8 h: number analyzed (Participants) | 6 | 6 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 4-8 h | 113.37 [10.10 to 205.00] | 344.17 [132.00 to 911.00] |  | 234.94 [97.70 to 473.00] | 603.40 [186.00 to 1100.00] |  | 417.33 [209.00 to 727.00]
  Unchanged ERT - 8-12 h: number analyzed (Participants) | 5 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 8-12 h | 54.95 [7.16 to 88.10] | 136.54 [21.70 to 198.00] |  | 88.86 [48.10 to 153.00] | 171.80 [137.00 to 217.00] |  | 113.88 [54.00 to 150.00]
  Unchanged ERT - 12-24 h: number analyzed (Participants) | 5 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 12-24 h | 43.04 [26.70 to 68.20] | 29.69 [9.35 to 72.20] |  | 65.46 [55.00 to 81.10] | 113.98 [85.60 to 159.00] |  | 96.03 [61.50 to 167.00]
  Unchanged ZID - 0-4 h: number analyzed (Participants) | 6 | 0 | 3 | 6 | 0 | 6 | 6
  Unchanged ZID - 0-4 h | 624.50 [383.00 to 824.00] |  | 1210.33 [691.00 to 1570.00] | 1465.00 [1465.00 to 1640.00] |  | 1855.00 [1090.00 to 2200.00] | 1870.00 [1320.00 to 2280.00]
  Unchanged ZID - 4-8 h: number analyzed (Participants) | 6 | 0 | 1 | 6 | 0 | 6 | 6
  Unchanged ZID - 4-8 h | 110.20 [7.22 to 173.00] |  | 302.00 [302.00 to 302.00] | 246.00 [219.00 to 307.00] |  | 556.83 [403.00 to 689.00] | 654.33 [253.00 to 1170.00]
  Unchanged ZID - 8-12 h: number analyzed (Participants) | 5 | 0 | 5 | 6 | 0 | 6 | 6
  Unchanged ZID - 8-12 h | 27.93 [3.55 to 45.10] |  | 45.58 [23.10 to 55.40] | 62.98 [40.20 to 93.60] |  | 175.00 [138.00 to 212.00] | 113.78 [27.70 to 160.00]
  Unchanged ZID - 12-24 h: number analyzed (Participants) | 5 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 12-24 h | 14.75 [7.36 to 25.40] |  | 62.37 [18.70 to 124.00] | 32.48 [13.30 to 44.80] |  | 67.67 [45.30 to 84.20] | 59.50 [34.00 to 85.60]

49. Secondary Outcome: Cumulative Amounts of Unchanged ERT and Unchanged ZID Excreted in Urine From Zero (Predose) to 24 h Following Dose 7 (Ae,Urine(0-24),SS)
Description: Mean and minimum/maximum of the cumulative amount of unchanged ERT and the cumulative amount of unchanged ZID excreted in urine from zero (predose) to 24 h following Dose 7, Ae,urine(0-24) (mg), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 7 (Day 7) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 7 infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: mg
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
mg
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT | 552.83 [325.00 to 778.00] | 1067.33 [340.00 to 1700.00] |  | 1166 [652.00 to 2200.00] | 1898.00 [1060.00 to 3000.00] |  | 1624.50 [887.00 to 2320.00]
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 1 | 6 | 0 | 6 | 6
  Unchanged ZID | 770.17 [495.00 to 1030.00] |  | 1080.00 [1080.00 to 1080.00] | 1808.33 [1580.00 to 1970.00] |  | 2656.67 [1770.00 to 2930.00] | 2700.00 [2200.00 to 3070.00]

50. Secondary Outcome: Fractions (%) of ERT and ZID Excreted Unchanged in Urine (fe,Urine) During Each Nominal Time Collection Interval Following Dose 7
Description: Mean and minimum/maximum of the fraction of ERT and the fraction of ZID excreted unchanged in urine, fe,urine (%), during 0-4 h, 4-8 h, 8-12 h, and 12-24 h following Dose 7 by dose group. These fe,urine parameters are calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 7 (Day 7) infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: % of dose excreted unchanged
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
% of dose excreted unchanged
  Unchanged ERT - 0-4 h: number analyzed (Participants) | 6 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 0-4 h | 35.78 [20.80 to 52.50] | 35.09 [1.97 to 63.30] |  | 38.94 [21.70 to 74.60] | 33.68 [21.80 to 51.00] |  | 33.28 [15.60 to 55.80]
  Unchanged ERT - 4-8 h: number analyzed (Participants) | 6 | 6 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 4-8 h | 11.34 [1.01 to 20.50] | 17.19 [6.62 to 45.50] |  | 11.72 [4.89 to 23.60] | 20.08 [6.19 to 36.50] |  | 13.91 [6.96 to 24.20]
  Unchanged ERT - 8-12 h: number analyzed (Participants) | 5 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 8-12 h | 5.50 [0.72 to 8.81] | 6.83 [1.08 to 9.91] |  | 4.45 [2.41 to 7.67] | 5.73 [4.57 to 7.23] |  | 3.80 [1.80 to 5.01]
  Unchanged ERT - 12-24 h: number analyzed (Participants) | 5 | 5 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT - 12-24 h | 4.30 [2.67 to 6.82] | 1.48 [0.47 to 3.61] |  | 3.27 [2.75 to 4.06] | 3.80 [2.85 to 5.30] |  | 3.20 [2.05 to 5.56]
  Unchanged ZID - 0-4 h: number analyzed (Participants) | 6 | 0 | 3 | 6 | 0 | 6 | 6
  Unchanged ZID - 0-4 h | 62.45 [38.30 to 82.40] |  | 60.40 [34.50 to 78.40] | 73.27 [62.60 to 82.10] |  | 61.85 [36.40 to 73.40] | 62.38 [44.00 to 76.00]
  Unchanged ZID - 4-8 h: number analyzed (Participants) | 6 | 0 | 1 | 6 | 0 | 6 | 6
  Unchanged ZID - 4-8 h | 11.02 [0.72 to 17.30] |  | 15.10 [15.10 to 15.10] | 12.28 [11.00 to 15.30] |  | 18.55 [13.40 to 23.00] | 21.84 [8.43 to 39.10]
  Unchanged ZID - 8-12 h: number analyzed (Participants) | 5 | 0 | 5 | 6 | 0 | 6 | 6
  Unchanged ZID - 8-12 h | 2.79 [0.36 to 4.51] |  | 2.28 [1.16 to 2.77] | 3.15 [2.01 to 4.68] |  | 5.84 [4.61 to 7.05] | 3.79 [0.92 to 5.34]
  Unchanged ZID - 12-24 h: number analyzed (Participants) | 5 | 0 | 6 | 6 | 0 | 6 | 6
  Unchanged ZID - 12-24 h | 1.48 [0.74 to 2.54] |  | 3.12 [0.93 to 6.20] | 1.63 [0.67 to 2.24] |  | 2.26 [1.51 to 2.81] | 1.98 [1.13 to 2.85]

51. Secondary Outcome: Fractions (%) of ERT and ZID Excreted Unchanged in Urine From Zero (Predose) to 24 h Following Dose 7 (fe,Urine(0-24),SS)
Description: Mean and minimum/maximum of the fraction of ERT and the fraction of ZID excreted unchanged in urine from zero (predose) to 24 h following Dose 7, fe,urine(0-24) (%), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 7 (Day 7) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 7 infusion
Population: as for outcome 11
Measure: Mean (Full Range); unit: % of dose excreted unchanged
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
% of dose excreted unchanged
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT | 55.28 [32.50 to 77.80] | 53.35 [17.00 to 84.90] |  | 58.36 [32.60 to 110.00] | 63.28 [35.50 to 100.00] |  | 54.20 [29.60 to 77.40]
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 1 | 6 | 0 | 6 | 6
  Unchanged ZID | 77.02 [49.50 to 103.00] |  | 53.80 [53.80 to 53.80] | 90.35 [78.80 to 98.50] |  | 88.48 [59.00 to 97.50] | 89.93 [73.30 to 102.00]

52. Secondary Outcome: Renal Clearance of ERT and ZID From Dosing Until the Last Collected Concentration for Dose 7 (CLR(0-24),SS)
Description: Geometric mean (GM), and coefficient of variation percentage (CV%) of renal clearance of ERT and ZID from dosing until the last collected concentration for Dose 7 (24 h postdose), CLR(0-24) (mL/h), by dose group. This parameter is calculated using a combination of Phoenix WinNonlin and SAS version 9.4 or above.
Time Frame: 0-1 h pre-start of Dose 7 (Day 7) infusion and 0-4 h, 4-8 h, 8-12 h, and 12-24 h post-start of Dose 7 infusion
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
L/h
  Unchanged ERT: number analyzed (Participants) | 6 | 6 | 0 | 5 | 5 | 0 | 6
  Unchanged ERT | 0.74 (28) | 0.78 (53) |  | 0.84 (48) | 0.92 (37) |  | 0.9 (44)
  Unchanged ZID: number analyzed (Participants) | 6 | 0 | 1 | 6 | 0 | 6 | 6
  Unchanged ZID | 5.59 (35) |  | 4.68 (NA) — Cannot be calculated as data only available for one participant | 5.84 (25) |  | 6.8 (25) | 6.77 (12)

ADVERSE EVENTS:
Time Frame: AEs were documented from the time of starting study drug administration through the time of Final Visit (Day 11 + 3 days)
Arm/Group | Cohort 1 - WCK 6777 2 g | Cohort 2 - ERT 2 g | Cohort 3 - ZID 2 g | Cohort 4 - WCK 6777 4 g | Cohort 5 - ERT 3 g | Cohort 6 - ZID 3 g | Cohort 7 - WCK 6777 6 g | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/6 | 5/6 | 4/6 | 2/6 | 4/6 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - WCK 6777 2 g (N=6) | Cohort 2 - ERT 2 g (N=6) | Cohort 3 - ZID 2 g (N=6) | Cohort 4 - WCK 6777 4 g (N=6) | Cohort 5 - ERT 3 g (N=6) | Cohort 6 - ZID 3 g (N=6) | Cohort 7 - WCK 6777 6 g (N=6) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 2 (5) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Infusion site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site papule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Injection site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05645757/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05645757/SAP_002.pdf
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT05645757/ICF_000.pdf